CLINICAL TRIAL: NCT03762434
Title: The Effectiveness of a Lifestyle Intervention Programme Using Mobile Application vs Booklet for Adult With Metabolic Syndrome _ a Pilot Study
Brief Title: Effectiveness of a Lifestyle Intervention Programme Using Mobile Application vs Booklet for Adult With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eliza Wong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1-BE0N
Record Dates: First submitted 2018-11-23; First posted 2018-12-03 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Metabolic Syndrome
Keywords: life style modification program; mobile application; metabolic sydrome; booklet; RCT
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: A multisite randomized controlled trial with two arms: MetS app group and , booklet group
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation and masking: A statistician will use computer-generated randomisation to determine random allocation. Eligible participants will be randomly allocated to either the control ( booklet group ) or the intervention group ( MetS app group) according to an allocation sequence prepared by the statistician before the start of the study. The patients will be randomised at a ratio of 1:1, with stratification by study site. Small cards indicating the group assignments will be placed in opaque sealed envelopes, which will be opened by the research assistant after each patient has completed the baseline questionnaires. In this study, the statisticians, outcome assessors and research assistant assigned to perform data input will be blinded to the allocation sequence. Given the type of intervention, however, the intervention group will be unmasked to the participants and the research nurse performing the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile app (Active Comparator): Mobile app: The participants will receive a Life style Modification Program with the support of mobile application (MetS app). The participants can view the similar knowledge content related to metabolic syndrome in their own smart phone. In addition, a membership area of the Mets app provides individual support of self- health monitoring, goal setting of exercise plan and exercise record. A user guide of the MetS app will be provided to the participants to take home after the app installment and briefing.
  Interventions: Other: mobile application
- booklet (Active Comparator): The participants will receive the Life Style Modification programme with the support of a Hong Kong version Metabolic Syndrome (MetS) booklet to take home and use for 3 months. The booklet had been modified from a booklet of a Life Style Intervention Programme (LIP) in China and the principal investigator of this proposal was the core team members of the previous project . The booklet content covers 26 pages about the metabolic syndrome and risk factors, suggested life style modification tips in terms of exercise, diet, smoking, mediation and stress management . The major component of the booklet for the change is the language translated from simplified Chinese to traditional Chinese and slight adjustment about the advice on vegetable choice due to difference in type of available vegetables in Hong Kong.
  Interventions: Other: mobile application

INTERVENTIONS:
Other: mobile application — Mobile app: The participants can view the Life style modification program by using the app. In addition, a membership area of the app provides individual support of self- health monitoring, goal setting of exercise plan and exercise record. A user guide of the MetS app will be provided to the participants to take home after the briefing.
  Booklet : The booklet content covers 26 pages about the metabolic syndrome and risk factors, suggested life style modification tips in terms of exercise, diet, smoking, mediation and stress management.
  Other Names: Booklet

SUMMARY:
Aims This Pilot study aims to develop and determine the feasibility and acceptability of a mobile application (MetS app) together with a modified Life style modification Program (LIP) for soon-to-aged adults with metabolic syndrome (MetS) and to determine the sample size for the main RCT. .

Methods A prospective randomized control trial design with process evaluation will be adopted. Inclusion criteria are those MetS participants, age 45 or above, able to use a smart phone. A total of eighty eligible participants will be recruited from 2-3 community Centres. Control group will receive standard care while intervention group will receive a MetS app. Standard care consists of a modified three-month lifestyle modification booklet, a 30 minutes educational session. The intervention group will receive a 30 minute education session plus MetS support, which will be guided by health belief model to support an individual self- monitoring and record of health measures (body weight, blood pressure, waist circumference) and physical exercise (goal setting of exercise and record) across three months. All information from the LIP booklet are also installed in the MetS platform as well. The primary outcomes will be waist measure and the total physical exercise (GSLTPAQ). The secondary outcomes included cardio-metabolic risk factors, cardiovascular endurance, self-efficacy for exercise (SEE) and stress level (PSS-10) and quality of Life (SF12). Data will be collected at baseline, one-month (T1) and three-month (T2). SPSS version 23 and Generalized Estimating equations (GEE) model will be employed to examine the effects of the LIP with MetS app support.

DETAILED DESCRIPTION:
Background Educational programme intervention on Lifestyle modification is recommended as the primary intervention for metabolic syndrome (MetS), a cluster of cardio-metabolic risk factors with a high prevalence rate globally and locally. Recent studies of lifestyle intervention program (LIP) have been reported as effective on physical indicators and quality of life (QoL) among MetS adult. However, they have the challenges in the delivery in making care scalable and little is known about the effect on exercise outcomes such as total exercise, cardiovascular endurance after exercise as well as whether the outcomes of this programme can be applied in Hong Kong and improved by adding the mobile application.

Aims This Pilot study aims to develop and determine the feasibility and acceptability of a mobile application (MetS app) together with a modified Life style modification Program (LIP) for soon-to-aged adults with metabolic syndrome (MetS) and to determine the sample size for the main RCT. .

Methods A prospective randomized control trial design with process evaluation will be adopted. Inclusion criteria are those MetS participants, age 45 or above, able to use a smart phone. A total of eighty eligible participants will be recruited from 2-3 community Centres. Control group will receive standard care while intervention group will receive a MetS app. Standard care consists of a modified three-month lifestyle modification booklet, a 30 minutes educational session. The intervention group will receive a 30 minute education session plus MetS support, which will be guided by health belief model to support an individual self- monitoring and record of health measures (body weight, blood pressure, waist circumference) and physical exercise (goal setting of exercise and record) across three months. All information from the LIP booklet are also installed in the MetS platform as well. The primary outcomes will be waist measure and the total physical exercise (GSLTPAQ). The secondary outcomes included cardio-metabolic risk factors, cardiovascular endurance, self-efficacy for exercise (SEE) and stress level (PSS-10) and quality of Life (SF12). Data will be collected at baseline, one-month (T1) and three-month (T2). SPSS version 23 and Generalized Estimating equations (GEE) model will be employed to examine the effects of the LIP with MetS app support.

Significance This pilot study will provide insights to guide the main study. The findings will facilitate the development of MetS app that could support the self-efficacy for physical health monitoring and exercise of patients with MetS. Such programme may enhance patient's self-management and monitoring of MetS, exercise behavior sustainability that will be beneficial to reduced MetS risk profile, and improves psychological health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants who satisfy the inclusion and exclusion criteria will be invited to participate in the RCT. The inclusion criteria are those :

  1. Ethnic Chinese Client who has a smart phone.
  2. Adult age 45 or over
  3. MetS Clients [1] with central obesity (male >90 cm , female > 80cm ) plus two items of the followings :

     * Raised triglycerides ≥ 150 mg/dL (1.7 mmol/L) or specific treatment for this lipid abnormality
     * Reduced HDL cholesterol < 40 mg/dL (1.03 mmol/L) in males < 50 mg/dL (1.29 mmol/L) in females or treatment for this lipid abnormality
     * Raised blood pressure systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg or treatment of previously diagnosed hypertension (HT)
     * Raised fasting plasma glucose (FPG) ≥ 100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes (DM)

Exclusion Criteria:

* Clients with physical, mental, visual, or cognitive impairments with regular medical follow-ups and treatment, and those who have musculoskeletal disorders or other disabling diseases that may limit the practice of walking exercise will be excluded.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 1 month and 3 months
  body weight weighted at the same scale by the research assistant (RA) in the follow up
Change in total physical exercise | baseline, 1 month and 3 months
  Total physical exercise quantified with a modified version of the GSLTPAQ [31-32]. The patients were instructed to indicate the amount of exercises and to rank the exercises in the order of difficulty (strenuous, moderate, and mild). Total physical exercise will be computed by summing up the total number of sessions per week multiplied by minutes per session. The scale has been widely used in empirical studies and it has been shown to have good psychometric properties with acceptable test-retest reliability (ranged from 0.62 to 0.81), and correlated with maximum oxygen consumption, treadmill time and other similar physical activity questionnaire. [31-32].

SECONDARY OUTCOMES:
Change in Chinese version of Self-Efficacy for Exercise (SEE-C) | baseline, 1 month and 3 months
  The SEE-C consists of nine items, and responses are made on a 0-10 scale. The sum of the responses to all nine items yields the final composite score ranging from 0-90. The C-SE has been proved to be reliable with good psychometric properties of Cronbach's alpha coefficient 0.75 for Taiwan Chinese older adults
change in Cardiovascular endurance test. | baseline, 3 mobnths
  it is a three -minute step test to test the cardiovascular functional endurance after exercise across the age span and gender. A participant step on and off of a 12 inch high bench / or stair for 3 minutes. Then pulse will be taken afterward while the participant remain standing. Compare the heart rate with the table according to the age and gender to determine the fitness in a range of 7 score from excellent, good, above average, average, below average, poor and very poor . Validity of this test has been established in previous studies. [35] .
Change in Perceived stress scale (PSS-10) | baseline, 1 month and 3 months
  Ten self-report items measure the degree to which situations in one's life are appraised as stressful and the current levels of experienced stress in the last month. Summative scores range from 0 to 40, with a higher score indicating higher stress level. These scores have been used as outcome measures of experienced levels of stress. The psychometric properties of the Chinese version of PSS-10 were satisfactory with Cronbach's alphas >0.75 in a local study for Chinese cardiac patients. [36]
Hospitalization frequency | baseline, 3 months
  Recent hospitalization frequency (number of hospitalization visit and hospitalization in last three month) will be asked by Research assistant (RA) at baseline and at 3 months.
Mets app usage frequency | monthly till 3 month
  MetS app usage (frequency per week) will be collected by RA by retrieving the data from the app server for the intervention group
Booklet usage frequency | baseline, 1 month and 3 months
  Booklet usage (frequency per week) will be collected for the control group at baseline, 1month and 3 months.
Waist circumference (cm) | baseline, 1 month and 3 months
  The Waist circumference is measured by a trained RA with a tape (cm) at the midpoint between the top of the iliac crest and the lower margin of the last rib in the standing position at the end of several consecutive natural breaths. Data will be collected at baseline, 1month and 3 months.
Blood pressure (mmHg) | baseline, 1month and 3 months.
  Systolic and diastolic blood pressure (mmHg) is measured by a trained RA using same equipment. Data will be collected at baseline, 1month and 3 months.
Lipid level (mmol/L) | baseline and 3 months
  Lipid level: A drop of blood sample will be taken by using a finger stick to measure LDL cholesterol (mmol/L), and HDL cholesterol (mmol/L), and triglycerides (mmol/L). The data can be analysed immediately by using auto-analyser and the participants are asked to have 8 hours fasting. Data will be collected by RA at baseline, 1month and 3 months.
Fasting blood glucose level (mmol/L) | baseline, 1 month and 3 months
  The participants are asked to have 8 hours fasting before blood taken. A drop of blood will be collected by finger stick by RA using same glucometer to measure the fasting blood glucose level at baseline, 1month and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Eliza ML Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Sai Kung community centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The result will be published .